CLINICAL TRIAL: NCT06136780
Title: Impact of Free Reading Glasses on Work and Visual Function Following Cataract Surgery in Honduras: The POWER Trial (Post-Operative Work-Related Effect of Reading Glasses)
Brief Title: Impact of Free Reading Glasses on Work and Visual Function Following Cataract Surgery in Honduras
Acronym: POWER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Advanced Center for Eyecare Global (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POWER Trial
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Free reading glasses immediately after cataract surgery
  Interventions: Other: Free reading glasses immediately following surgery
- Control (No Intervention): Free reading glasses will be given 4 months after cataract surgery

INTERVENTIONS:
Other: Free reading glasses immediately following surgery — Free reading glasses will be given immediately after cataract surgery in the intervention arm and four months after cataract surgery in the control arm.
  Arms: Experimental

SUMMARY:
Cataract surgery improves vision and is therefore assumed to improve a person's ability to work and function. Following cataract surgery, most patients do not need glasses to see clearly at distance, but they do require glasses to see clearly up close. If a patient is unable to acquire reading glasses after surgery due to either financial or logistical reasons, their ability to resume work and functioning may be compromised, diminishing the overall benefit to be gained from cataract surgery. Patients in the developing world may be affected disproportionately due to difficulty accessing care postoperatively. In this study, patients receiving cataract surgery at a clinic in Comayagua, Honduras will be randomized to either receive free reading glasses immediately after surgery or four months later. The primary outcome is the proportion of subjects who report that vision interferes with their ability to work. Secondary outcomes will include the number of hours worked each week at productive activities, income level, and visual functioning. The hypotheses are that the patients who receive free reading glasses immediately following surgery will be less likely to report that their vision interferes with their ability to work, they will work at productive activities a greater number of hours each week, their incomes will be higher, and their visual function scores will be higher.

DETAILED DESCRIPTION:
Introduction The goal of cataract surgery is to improve a patient's vision and by extension, their ability to work and function. Cataract is the clouding of the lens of the eye, and during cataract surgery, the ophthalmologist removes the clouded lens and replaces it with a manufactured lens. Both the natural and the manufactured lens focus light onto the retina, and the length and shape of the eye determine what power intraocular lens to insert at the time of surgery. Using measures taken prior to surgery, cataract surgeons aim to provide patients with clear vision at a distance without glasses. The surgery, when done with the most widely available intraocular lenses by this approach, typically leaves a patient in focus at a distance and dependent on glasses for near work. The assumption with this approach is that the improved vision will enable the patient to return to work and normal functioning. However, in a recent study in Comayagua, Honduras at a facility that exclusively serves low-resource communities (working paper), 75% of patients reported that their vision still interfered with their ability to work four months after cataract surgery. A much smaller number would be expected if cataract surgery alone were able to restore good, functional vision.

A possible explanation for the persistence of vision problems that interfere with work in this cohort is the need for reading glasses. Many occupations involve near work, and having glasses specifically for near work has been shown to increase productivity. Good near vision is also required for a wide variety of tasks around the home and for attending to basic life needs such as dressing and eating. Ideally, following cataract surgery, patients are tested for prescription glasses around one month post-operatively, and glasses prescriptions are written at that time. Postoperative visits and care for cataract patients in the developing world often does not meet this ideal. Returning to the clinic after cataract surgery for postoperative visits can be difficult or impossible, and though they are instructed to return to the clinic to be seen, many patients are lost to follow-up. For the patients who are able to return to be checked, glasses prescriptions are written if they are needed, but such prescriptions are often expensive to fill. Therefore, many patients do not receive any spectacle correction following cataract surgery in the developing world. This is in spite of the fact that the vast majority of these patients at least need glasses for near work.

In a follow-up study to address the effect of reading glasses on work following cataract surgery, 68 patients in the same clinic in Comayagua, Honduras were given free reading glasses at the time of cataract surgery. Three months later, only 22% (n=11) of the 51 patients contacted reported that their vision interfered with their ability to work, and 78%(n=40) reported that the reading glasses that they were given made it easier to work.

Obtaining glasses following surgery might involve significant barriers, including economics (patients are unable to afford the glasses that they need), logistics (patients are unable to travel to a pharmacy that carries glasses) or information (patients lack an understanding of the need for and utility of reading glasses after surgery). Distributing very low-cost reading glasses (~$0.60/pair) at the time of cataract surgery could potentially address these problems. For minimal cost and with few logistical hurdles, giving free reading glasses to postoperative cataract patients ensures that all patients, at a minimum, receive some assistance with near vision. Patients would still be encouraged to follow-up for a custom pair of prescription glasses, as this approach will not address all postoperative need for glasses. However, even if complete follow-up care is inaccessible to a patient for financial or logistical reasons, distribution of free reading glasses at the time of surgery could increase the odds that a person has functional near vision after surgery.

In this study, we want to directly test the effect of providing free reading glasses following cataract surgery on work, income, and functioning through a randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataracts causing VA <6/12 OU, scheduled for cataract surgery at San Benito Jose Clinic in Comayagua Honduras during the week of 3.17.2024 - 3.23.2024.
* Age 50 or older.

Exclusion Criteria:

* Previous eye surgery. Ocular comorbidities. Cataract surgery complications resulting in aphakia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-17 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that reports vision interferes with ability to work | Four months after cataract surgery
  Percentage of total

SECONDARY OUTCOMES:
Number of hours per week engaged in productive activities | Four months after cataract surgery
  Productive activities including paid work, unpaid work for self, unpaid work in household
Paid monthly income | Four months after cataract surgery
  Categorical variable
Visual function score based on National Eye Institute's Visual Function Questionnaire-8. | Four months after cataract surgery
  Continuous variable generated from validated iinstrument

CONTACTS AND LOCATIONS:
Overall Officials: Sara OConnor, MD, MPH, Principal Investigator — Advanced Center for Eyecare Global

IPD SHARING:
Plan to Share IPD: Yes
All data other than personal ID's will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: https://acecaresglobal.org/